CLINICAL TRIAL: NCT02221960
Title: A Phase 1 Multicenter, Open-label, Dose-escalation and Dose-expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Antitumor Activity of MEDI6383 Alone and in Combination With MEDI4736 in Adult Subjects With Select Advanced Solid Tumors
Brief Title: A Phase 1 Study to Evaluate MEDI6383 Alone and in Combination With MEDI4736 in Adult Subjects With Select Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6050C00001
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Recurrent or Metastatic Solid Tumors
Keywords: Recurrent or metastatic solid tumors, MEDI6383, OX40
MeSH Terms: conditions — Recurrence | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monotherapy Arm (Experimental): MEDI6383
  Interventions: Biological: MEDI6383
- Combination Arm (Experimental): MEDI6383 and MEDI4736
  Interventions: Biological: MEDI6383 and MEDI4736

INTERVENTIONS:
Biological: MEDI6383 — Subjects will receive MEDI6383 until disease progression or adverse event.
  Arms: Monotherapy Arm
Biological: MEDI6383 and MEDI4736 — Subjects will recieve MEDI6383 and MEDI4736 until disease progression or adverse event.
  Arms: Combination Arm

SUMMARY:
To evaluate MEDI6383 when given alone or together with MEDI4736 in adult subjects with recurrent or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open-label, dose-escalation, and dose-expansion study to evaluate the safety, tolerability, pharmacokinetics, immunogenicity, pharmacodynamics, and antitumor activity of MEDI6383 alone and in combination with MEDI4736 in adult subjects with recurrent or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects; age ≥ 18
2. Written informed consent must be obtained
3. Subjects must meet the following criteria:

   1. Have recurrent or metastatic solid tumors
   2. Must have received and have progressed, are refractory, or are intolerant to standard therapy appropriate for the specific tumor type. Subjects should not have received more than 5 prior lines of therapy for recurrent or metastatic disease including both standards of care and investigational therapies
4. Subjects must have at least 1 lesion
5. Subjects must consent to provide archived tumor specimens and / or tumor biopsy for correlative biomarker studies.
6. Eastern Cooperative Oncology Group performance score of 0 or 1
7. In the opinion of the invesgator likely to complete ≥ 8 weeks of treatment.
8. Adequate organ function as determined by:

   i. Absolute neutrophil count ≥ 1.5 x 109/L (1,500/mm3) ii.Platelet count ≥ 100 x 109/L (100,000/mm3) iii.Hemoglobin ≥ 9.0 g/dL within first 2 weeks prior to first dose of investigational product iv.Calculated creatinine clearance* (CrCl) or 24 hour urine CrCl > 50 mL/min v.Total bilirubin ≤ 1.5× ULN; for subjects with documented/suspected Gilbert's disease, bilirubin ≤ 3× ULN vi.Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5× ULN vii.Serum Electrolytes within normal limits
9. Females of childbearing potential who are sexually active with a nonsterilized male partner must use 2 methods of highly effective contraception from screening, and must agree to continue using such precautions for 90 days after the final dose of investigational product; 10) Nonsterilized males who are sexually active with a female partner of childbearing potential must use a highly effective method of contraception from Day 1 through 90 days after receipt of the final dose of investigational product

Exclusion Criteria:

1. Prior treatment with TNFRSF agonists including OX40, CD27, CD137 (4-1BB), CD357 (GITR) .
2. Subjects who have received prior therapy with regimens containing CTLA-4, PDL-1, or PD-1 antagonists are NOT permitted to enroll unless all of the following apply:

   * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy
   * All AEs while receiving prior immunotherapy must have resolved to ≤ Grade 1 or baseline prior to screening for this study.
3. Must not have experienced a ≥ Grade 3 AE or neurologic or ocular AE of any grade while receiving prior immunotherapy
4. History of severe allergic reactions to any unknown allergens or any components of the study drug formulations
5. Active or prior documented autoimmune disease within the past 2 years.
6. Untreated central nervous system metastatic disease l
7. Concurrent enrollment in another clinical study, unless it is an observational (non interventional) clinical study or the follow-up period of an interventional study
8. Receipt of anticancer therapy within 28 days prior to the first dose of Investigational Product
9. Any concurrent chemotherapy, immunotherapy, or biologic or hormonal therapy for cancer treatment.
10. Unresolved toxicities from prior anticancer therapy
11. Systemic anticoagulation or daily aspirin dose exceeding 325 mg per day
12. Current or prior use of immunosuppressive medication within 14 days prior to the first dose of MEDI6383. )
13. History of primary immunodeficiency, solid organ transplantation, or tuberculosis
14. True positive test results for human immunodeficiency virus (HIV) or hepatitis B or C
15. Receipt of live, attenuated vaccine within 28 days prior to the first dose of investigational products )
16. Pregnant or breastfeeding women
17. Major surgery (as defined by the investigator) within 4 weeks prior to first dose of MEDI6383 or still recovering from prior surgery. Local surgery of isolated lesions for palliative intent is acceptable
18. Other invasive malignancy within 2 years

    -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Safety | From time of informed consent through 12 weeks after last dose of investigational product
  Primary endpoint will be the number (%) of subjects with adverse events and serious adverse events.

SECONDARY OUTCOMES:
Preliminary Antitumor Activity | Duration of Study
  The endpoints for assessment of antitumor activity include objective response (OR), disease control (DC), duration of response (DoR), progression-free survival (PFS), and 3-year overall survival (OS)
Pharmacokinetics of MEDI6383 or MEDI6383/MEDI4736 | From time of informed consent through 12 weeks after last dose of investigational product
  When MEDI6383 is administered alone, the endpoints for assessment of PK of MEDI6383 include individual subject MEDI6383 concentrations in serum at different time points after MEDI6383 administration. When MEDI6383 is administered together with MEDI4736, the endpoints for assessment of PK of MEDI6383 and MEDI4736 include individual subject MEDI6383 and MEDI4736 concentrations in serum at different time points after MEDI6383 and MEDI4736 administration. PK Parameters that may be modeled may include Cmax, Area Under the concentration-time curve, Clearance, and terminal half-live.
Biomarker Activity | From time of informed consent through 12 weeks after last dose of investigational product
  The endpoints for assessment of pharmacodynamic activity include immunohistochemistry of tumor biopsies and assessment of tumor-infiltrating lymphocyte phenotypic markers
Immunogenicity | From time of informed consent through 12 weeks after last dose of investigational product
  The endpoint for for the assessment of immunogenicity will include the number and percentage of subjects that develop anti-drug antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Medimmune Medimmune, Study Director — MedImmune LLC
Locations (8):
- United States (7):
  - Research Site, La Jolla, California
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Chicago, Illinois
  - Research Site, New York, New York
  - Research Site, Portland, Oregon
  - Research Site, Nashville, Tennessee
- Research Site, Parkville, Australia